CLINICAL TRIAL: NCT01265394
Title: A Single-arm, Open-label, Multi-center Study to Determine the Specificity of Flutemetamol (18F) Injection for Excluding the Presence of Brain Amyloid in Healthy Young Adult Subjects Aged 18 to 40
Brief Title: Positron Emission Tomography (PET) Amyloid Imaging of the Brain in Healthy Young Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-067-015
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Amyloid; Magnetic resonance imaging; Positron Emission Tomography; Standard uptake value ratios; Healthy Subjects
MeSH Terms: conditions — Alzheimer Disease | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (18F) Flutemetamol (Experimental)
  Interventions: Drug: [18F] Flutemetamol

INTERVENTIONS:
Drug: [18F] Flutemetamol — Flutemetamol (18F) Injection, 185 MBq/5 mCi, single intravenous injection.
  Other Names: AH110690

SUMMARY:
Amyloid is an abnormal chemical found in the brain of patients with Alzheimer's Disease (AD). The study drug helps produce pictures of amyloid in the brain. The purpose of this study is to determine how well the study drug performs in young healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject age is 18 to 40 years.
* The subject has no evidence of thinking or memory problems by medical history.
* The subject has a normal MRI scan.
* The subject's general health is adequate to comply with study procedures.
* The subject is willing and able to participate in all study procedures.

Exclusion Criteria:

* The subject has received any medical ionizing radiation exposure in the last 12 months (except planar x-ray or head CT).
* The subject has a contraindication for (cannot undergo) MRI.
* The subject has a history of head injury with loss of consciousness.
* The subject has any significant medical, psychiatric or neurological condition that might be associated with brain pathology.
* The subject has a family history of Alzheimer's Disease (AD); more than 1 first-degree relative.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, MD, PhD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- (18F) Flutemetamol: [18F] Flutemetamol : Flutemetamol (18F) Injection, 185 MBq/5 mCi, single intravenous injection.
Period: Overall Study
Arm/Group | (18F) Flutemetamol
Started | 218
Completed | 181
Not Completed | 37
Not completed — Subjects withdrawn | 37

BASELINE CHARACTERISTICS:
Population: This is the number of participants that completed.
Arm/Group | (18F) Flutemetamol
Number analyzed (Participants) | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 181
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 78
Region of Enrollment [Number; unit: participants]
  United States | 127
  Belgium | 10
  Finland | 19
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Brain Scans in Healthy Young Adults Subjects Which do Not Show Amyloid
Description: The visual assessment of Flutemetamol PET image was performed by independent readers trained in the evaluation of PET brain amyloid imaging.
  The measure would consisted of the number of brain scans with amyloid (abnormal reading) or without amyloid (normal reading).
Time Frame: PET scans performed on patients 90 minutes post Flutemetmol Administration
Population: Healthy young adult subjects aged 18 to 40 are presumed to be amyloid negative
Measure: Number; unit: Brain Scans Read
Groups:
- Normal and Abnormal Reads With or Without Amyloid: Each Subject received a dose of [18F] Flutemetamol : Flutemetamol (18F) Injection, 185 MBq/5 mCi, single intravenous injection.
Arm/Group | Normal and Abnormal Reads With or Without Amyloid
Number analyzed (Participants) | 181
Brain Scans Read
  Reader 1 -Normal Read-no amyloid | 181 [98.0 to 100.0]
  Reader 1- Abnormal Read- amyloid is present | 0 [60.6 to 74.7]
  Reader 2 - Normal Read-no amyloid | 123 [97.0 to 100.0]
  Reader 2 - Abnormal Read-amyloid is present | 58 [97.0 to 100.0]
  Reader 3 - Normal Read-no amyloid | 180 [96.1 to 99.9]
  Reader 3 - Abnormal Read-amyloid is present | 1
  Reader 4 - Normal Read-no amyloid | 180
  Reader 4 - Abnormal Read-amyloid is present | 1
  Reader 5 - Normal Read-no amyloid | 179
  Reader 5 - Abnormal Read-amyloid is present | 2

2. Secondary Outcome: Measurement of Amyloid Content in Different Parts of the Brain
Description: Is the computerized measurement of amyloid content in different parts of the brain.
  The Standard Uptake Value Ratio (SUVR) is defined as an average of frontal, anterior cingulate, pariteal, lateral-temporal and posterior cingulate / precuneous uptake following administration of Flutemetamol F18 Injection.
  The Standard Uptake Value Ratio is calculated for two regions of the brain, the Cerebullum and the Pons regions.
  The Standard Uptake Value Ratio is calculated for two regions of the brain, the Cerebullum and the Pons regions. Both regions of the brain will provide the SUVR measurements.
Time Frame: PET scans performed on patients 90 minutes post Flutemetmol Administration
Population: The Standard Uptake Value Ratio is calculated for two regions of the brain, the Cerebullum and the Pons regions. Both regions of the brain will provide the SUVR measurements.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value Ratio ( SUVR)
Groups:
- (18F) Flutemetamol Injection: Flutemetamol (18F) Injection, 185 MBq/5 mCi, single intravenous injection.
Arm/Group | (18F) Flutemetamol Injection
Number analyzed (Participants) | 181
Standard Uptake Value Ratio ( SUVR)
  Cerebullum Region | 1.12 (0.097) [1.108 to 1.136]
  Pons Region | 0.49 (0.036) [0.487 to 0.498]

ADVERSE EVENTS:
Arm/Group | (18F) Flutemetamol
Serious Adverse Events (participants affected / at risk) | 0/181
Other Adverse Events (participants affected / at risk) | 27/181
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (18F) Flutemetamol (N=181)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (9)
General Disorders and Administration Site Conditions (General disorders) | 12 (12)
Vascular System Disorders (Vascular disorders) | 11 (11)
Vascular System Disorders-Flushing (Vascular disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No